CLINICAL TRIAL: NCT01395043
Title: TAP-catheter With Intermittent Bolus Injections of Bupivacain, an Alternative to Epidural Catheter Infusion After Colon Surgery?
Brief Title: Transversus Abdominis Plane Catheter: a Study of Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Nils Bjerregaard, Departement of anesthesia, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N-20100001
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-01

CONDITIONS: Postoperative Pain
Keywords: Transversus Abdominis Plane catheter; TAP catheter
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAP-catheter (Other): Each patient receives bilateral TAP-catheters preoperatively.
  Interventions: Procedure: Placing bilateral TAP-catheters preoperatively; Drug: Bupivacain 2.5 mg/ml with epinephrine bolus in TAP-catheters

INTERVENTIONS:
Procedure: Placing bilateral TAP-catheters preoperatively — Place bilateral TAP-catheters preoperatively and give repeated boluses of local analgetics in order to treat postoperative pain after colon-surgery.
  Other Names: Bilateral TAP-catheter
Drug: Bupivacain 2.5 mg/ml with epinephrine bolus in TAP-catheters — Intermittent boluses of Bupivacain 2.5 mg/ml with epinephrine, 20 ml in each catheter every 12 hours for the first 2 postoperative days.

SUMMARY:
Major abdominal surgery is associated with postoperative pain. Transversus Abdominis Plane(TAP) block has been shown to reduce pain and opioid-requirements after abdominal surgery. However a single block has a short effect of up to 12 hours depending on the type local-anesthetics used.

With this study we wish to investigate the possibilities to place a TAP-catheter in order to prolong the the effect of the TAP-block by giving repeatedly bolus-injections in the TAP catheter and to study the pain and the opioid requirements of patients undergoing elective colon-resection when given a TAP-catheter preoperatively.

Our hypothesis is that it is practical and technical possible to place bilateral TAP-catheters pre-operatively and that pain and opioid-requirements will be low.

DETAILED DESCRIPTION:
Postoperative pain is a major challenge in the work of anesthesia. Epidural catheter is the golden standard for postoperative pain management after major abdominal surgery. However a number of patient have absolute or relative contraindication to the placement of an epidural catheter. It is therefore necessary to find a good alternative to epidural catheter.

Transversus abdominis plane(TAP) block has been shown to provide analgesia of the abdominal wall and reduce opioid-requirements and pain after abdominal surgery.

However the effect of a TAP block is limited to the time of efficacy of the local analgesic used. Placing a TAP-catheter in order to prolong the effect of the TAP-block by repeatedly bolus-injections in the TAP-catheters has only been sporadically described and so far never investigated in a systematic way.

We will investigate the practical and technical possibility to place bilateral ultrasound-guided TAP-catheters pre-operatively on patients undergoing elective colon-resection. Further more we will evaluate the pain and opioid-requirement postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* elective open colon-resection
* adult
* written and informed consent

Exclusion Criteria:

* re-operation within the first 48 hours
* need for sedation and ventilator-support postoperatively
* accidental removal of catheter within the first 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Rasmussen, PhD, Study Chair — departement of anesthesiology, Aalborg Hospital
Locations (1):
- departement of anesthesiology, Aalborg University Hospital, Aalborg, North Denmark, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilateral Ultrasoundguide TAP-catheter: All patients receive bilateral ultrasound guided TAP-catheter and bolus injections of bupivacain 2.5 mg/mL with epinephrin 5 µg/mL every 12 hours in both catheters
Period: Overall Study
Arm/Group | Bilateral Ultrasoundguide TAP-catheter
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bilateral Ultrasoundguide TAP-catheter
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Region of Enrollment [Number; unit: participants]
  Denmark | 15

OUTCOME MEASURES:

1. Secondary Outcome: Opioid Requirements Postoperative
Description: Supplementary opioid requirements for the first 48 hours from arriving in the post anesthesia care unit. Results are total opioid-requirements for the first 48 hours. Way of administration was intravenous in all but 6 administrations. If given orally, a 1:3 ratio was used for conversion from oral to intravenous morphine.
Time Frame: 48 hours from arriving in the post anesthesia care unit.
Measure: Mean (95% Confidence Interval); unit: mg iv morphin equivalent
Groups:
- Bilateral Ultrasoundguide TAP-catheter: All patients receive bilateral ultrasound guided TAP-catheter and bolus injections of bupivacain 2,5 mg/mL with epinephrin 5 µg/mL every 12 hours in both catheters
Arm/Group | Bilateral Ultrasoundguide TAP-catheter
Number analyzed (Participants) | 15
mg iv morphin equivalent | 35 [22 to 39]

2. Primary Outcome: Postoperative Pain Using Numerical Rating Scale (NRS) 0-10
Description: NRS is a pain score and the score can vary between 0 and 10 by which 0 means no pain and 10 equals the worst possible pain.
  NRS was evaluated at the time 0, 1, 2, 4, 8 , 12, 18 , 24 and 36 hours after arriving in the post anesthesia care unit at rest and during coughing.
Time Frame: 0-36 hours postoperative
Measure: Median (Inter-Quartile Range); unit: Units on Numerical Rating Score
Arm/Group | Bilateral Ultrasoundguide TAP-catheter
Number analyzed (Participants) | 15
Units on Numerical Rating Score
  NRS at rest, all times | 3 [2 to 6]
  Overall NRS when coughing, all times | 5 [2 to 6]

ADVERSE EVENTS:
Arm/Group | Bilateral Ultrasoundguide TAP-catheter
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Not randomised or blinded. Limited number of patients. Dermatome level of the block and the incidence of postoperative nausea and vomiting was not registered. The study does not compare TAP-catheter and epidural catheter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes